CLINICAL TRIAL: NCT04689932
Title: Triferic AVNU Infusion Via Freedom Pump During Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rockwell Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RMFPC-ISS002
Record Dates: First submitted 2020-12-28; First posted 2020-12-30 (Actual); Results first posted 2022-01-18 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pre- Dialyzer Infusion and Post- Dialyzer Infusion (Experimental): On study day 1, day 3 and day 5, patients will receive 6.75 mg Fe/4.5 mL Triferic AVNU intravenously using the Freedom Pump-20 during hemodialysis into the pre-dialyzer blood line. On study day 2, day 4 and day 6, patients will receive the 6.75 mg Fe/4.5 mL Triferic AVNU intravenously using the Freedom Pump-20 during hemodialysis into the post dialysis blood line.
  Interventions: Drug: Triferic AVNU

INTERVENTIONS:
Drug: Triferic AVNU — Ferric Pyrophosphate Citrate
  Other Names: FPC

SUMMARY:
The main purpose of this study is to evaluate the delivery of Triferic AVNU intravenously using the Freedom Pump-20 during hemodialysis into the pre-dialyzer and post-dialyzer blood lines.

DETAILED DESCRIPTION:
This is a single center, multi dose, open label study assessing the delivery of Triferic AVNU administered intravenously to adult patients (> or equal to 18 years of age) using the Freedom Pump-20 during hemodialysis into the pre-dialyzer and post-dialyzer blood lines.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 years of age inclusive, at the time of signing the informed consent.
2. Receiving chronic hemodialysis for 3-4 hours each session 3x/week.
3. Medically stable according to the investigator opinion
4. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Hemodynamically unstable during hemodialysis
2. Evidence of active bleeding from the GI tract.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-06-19 (Actual); Study Completion 2021-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond D Pratt, MD, FACP, Study Director — Rockwell Medical
Locations (1):
- Luxury Dialysis, Webster, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pre- Dialyzer Infusion and Post- Dialyzer Infusion
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pre- Dialyzer Infusion and Post- Dialyzer Infusion
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 3
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Time for Complete Infusion of 4.5 mL Triferic AVNU Pre-Dialyzer
Description: The syringe pump and flow restrictor tubing has a nominal flow rate of 2 mL/hour. When the tubing is connected to the pre-dialyzer or post dialyzer blood circuit the administration time will vary due to the pressure in the dialyzer blood lines. For a 4.5 mL volume the target administration rate is 2.25 hours. The Product labeling for Triferic AVNU advises the dose (4.5 mL) to be administered over 3 to 4 hours.
Time Frame: On Days 1, 3, and 5, up to 3 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Pre- Dialyzer Infusion and Post- Dialyzer Infusion
Number analyzed (Participants) | 12
hours | 1.7 (2.0)

2. Primary Outcome: Time for Complete Infusion of 4.5 mL Triferic AVNU Post-Dialyzer
Description: as for outcome 1
Time Frame: On Days 2, 4, and 6, up to 3 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Pre- Dialyzer Infusion and Post- Dialyzer Infusion
Number analyzed (Participants) | 12
hours | 2.5 (2.8)

3. Secondary Outcome: Mean TSAT Max Pre-Dialyzer
Description: The maximum Transferrin saturation (TSATmax) for the infusion of FPC into the pre-dialyzer blood line when compared to the TSATmax when FPC is infused into the post-dialyzer blood line is an index of any loss of FPC during transit through the dialyzer (artificial kidney
Time Frame: up to 3 hours
Measure: Mean (Standard Deviation); unit: percentage of saturation
Arm/Group | Pre- Dialyzer Infusion and Post- Dialyzer Infusion
Number analyzed (Participants) | 12
percentage of saturation | 88 (101)

4. Secondary Outcome: Mean TSAT Max Post-Dialyzer
Description: as for outcome 3
Time Frame: up to 3 hours
Measure: Mean (Standard Deviation); unit: percentage of saturation
Arm/Group | Pre- Dialyzer Infusion and Post- Dialyzer Infusion
Number analyzed (Participants) | 12
percentage of saturation | 67 (81)

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Pre- Dialyzer Infusion: On study day 1, day 3 and day 5, patients will receive 6.75 mg Fe/4.5 mL Triferic AVNU intravenously using the Freedom Pump-20 during hemodialysis into the pre-dialyzer blood line.
  Triferic AVNU: Ferric Pyrophosphate Citrate
- Post- Dialyzer Infusion: On study day 2, day 4 and day 6, patients will receive the 6.75 mg Fe/4.5 mL Triferic AVNU intravenously using the Freedom Pump-20 during hemodialysis into the post dialysis blood line.
  Triferic AVNU: Ferric Pyrophosphate Citrate
Arm/Group | Pre- Dialyzer Infusion | Post- Dialyzer Infusion
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT04689932/Prot_SAP_000.pdf